CLINICAL TRIAL: NCT05596162
Title: The Effect of Low-Intensity Blood Flow Restriction Therapy on the Management of Acute Ankle Sprains
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No support
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eric N. Bowman, Assistant Professor of Orthopaedic Surgery, Division of Sports Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220838
Record Dates: First submitted 2022-10-16; First posted 2022-10-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree; Musculoskeletal Injury
Keywords: blood flow restriction; ankle sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be aware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction Group (Experimental): 1. Patient specific tourniquet settings to achieve 80% occlusion.
  2. Weight- 20% of 1 rep max, 4 sets 30-15-15-15 reps with 30 second rests between sets
  3. Exercises: The first phase will focus on active and passive range of motion of the ankle as well as non-weighted concentric exercises. Phase two will progress with gastrocnemius and soleus stretches along with body weight and light resistance band concentric and eccentric exercises focusing on posterior, anterior and lateral muscle groups of the lower limb. Phase three will introduce weighted, dynamic and proprioceptive exercises.
  Interventions: Other: Blood Flow Restriction Therapy
- Non-Blood Flow Restriction Group (Active Comparator): This group will perform the same exercises for the same volume without the use of BFR.
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: Blood Flow Restriction Therapy — Exercise with Blood Flow Restriction
  Arms: Blood Flow Restriction Group
Other: Standard Physical Therapy — Exercise without Blood Flow Restriction
  Arms: Non-Blood Flow Restriction Group

SUMMARY:
The primary objective of this study is to evaluate the feasibility of implementing BFR in the rehabilitation treatment of isolated ankle sprains as well as to evaluate the clinical benefits of BFR when compared to standard treatment. This study will evaluate the efficacy of using BFR therapy for the treatment of acute grade I and II ankle sprains. The investigators will evaluate clinical outcomes of range of motion (ROM) and strength testing of ankle dorsiflexion, plantarflexion, inversion, and eversion.

This will be a small, randomized control trial study. The investigators will enroll a total of 40 participants, 20 participants will undergo standard physical therapy for isolated lateral ankle sprains and 20 participants will undergo BFR therapy for an isolated lateral ankle sprain. Patients will be randomized into control and experimental group via block randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients will include English speaking student athletes aged 18 and older with clinical diagnosis of an isolated grade I or II lateral ankle sprain

Exclusion Criteria:

* History of DVT/PE, clotting disordered, peripheral arterial disease, hypertension (BP>140/90), coronary artery disease, or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time to Return to Play | From Time of Injury to 8 weeks after Injury
  Time from injury to to when injured ankle regains 90% plantarflexion strength compared to uninjured/contralateral side, using a dynamometer.

SECONDARY OUTCOMES:
Pain Level | Initial visit & 1, 2, 4, and 8 weeks after the initial visit
  Pain will be assessed with the Visual Analog Pain Scale (VAS). The minimum and maximum scores are 0 and 10 respectively with higher scores meaning a worse outcome.
Range of Motion | Initial visit & 1, 2, 4, and 8 weeks after the initial visit
  Range of motion of ankle dorsiflexion, plantarflexion, inversion, and eversion. It will be measured from 0 to 360 with higher scores meaning a worse outcome.
Strength Testing | Initial visit & 1, 2, 4, and 8 weeks after the initial visit
  Strength testing of ankle dorsiflexion, plantarflexion, inversion, and eversion. It will be measured from 0 to 5 with higher scores meaning a better outcome.
The Foot and Ankle Ability Measure (FAAM) Patient-Reported Score | Initial visit & 1, 2, 4, and 8 weeks after the initial visit
  The Foot and Ankle Ability Measure (FAAM) will be used to measure self-reported physical function. It will be measured from 0 to 116 with higher scores meaning a better outcome.
Foot and Ankle Outcome Score (FAOS) Patient-Reported Score | Initial visit & 1, 2, 4, and 8 weeks after the initial visit
  The Foot and Ankle Outcome Score (FAOS) will be used to measure self-reported physical function. It will be measured from 0 to 100% with higher scores meaning a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- VUMC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No